CLINICAL TRIAL: NCT06270147
Title: Single Blind Clinical Trial: Optimizing TAP Block Timing for Bariatric Surgery
Brief Title: Timing of TAP Blocks in Bariatric Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 16935
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early TAP block (Experimental): Patients in this group will receive TAP blocks at the beginning of the procedure
  Interventions: Drug: Bupivacaine-epinephrine
- Late TAP block (Active Comparator): Patients in this group will receive TAP blocks at the end of their procedure, which is the current standard practice.
  Interventions: Drug: Bupivacaine-epinephrine

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — A total of 60ml of 0.25% Bupivacaine with Epinephrine, divided into 4 aliquots, will be administered laparoscopically at two locations per side along the anterior axillary line between the costal margin and the iliac crest. TAP block timing will be disclosed to the operating surgeon to ensure the correct solution is administered at the appropriate time.

SUMMARY:
This clinical trial aims to determine the optimal timing for administering a Transversus Abdominis Plane (TAP) block in bariatric surgery, specifically investigating whether initiating TAP blocks at the beginning of surgery is more beneficial than at the end, which is the current practice. The study targets obese patients undergoing bariatric surgery, with a focus on reducing postoperative pain and opioid use. Key outcomes include recovery duration, pain levels, opioid consumption, and respiratory function. Successful results could establish early TAP block initiation as a standard practice, offering faster recovery, decreased opioid reliance, and reduced healthcare costs.

DETAILED DESCRIPTION:
Post-operative pain remains a critical aspect of patients' recovery, with approximately 70% of patients who undergo surgery reporting moderate to severe levels of pain post-operatively. Increased post-operative pain has adverse effects on psychological and physiological function including cardiovascular, respiratory, gastrointestinal, immune function and wound healing. In an era where patient centered care is at its peak and healthcare resources are limited, adequate post-operative pain management is crucial. It facilitates early mobilization, reduces the length of stay in hospital and overall costs on the healthcare system.

The transversus abdominis plane (TAP) block, a peripheral nerve block, has been shown to significantly reduce postoperative opioid requirements, even in the context of minimally invasive surgery (MIS). Furthermore, the literature clearly indicates the benefit of TAP blocks on post-operative analgesia in patients undergoing bariatric surgery. However, evidence regarding the ideal timing of TAP block administration in the bariatric population is lacking. In current practice, TAP blocks are generally administered after the surgery, and occasionally after induction of anesthesia. However emerging studies suggest that administering TAP blocks at the beginning of a procedure may result in superior recovery and pain control in the immediate period following open and laparoscopic surgery compared to at the end of a procedure.

The purpose of the study is to assess the timing of TAP block administration in bariatric surgery patients on the immediate post-operative recovery period. This will be determined by the amount opioids required in the post-anesthetic recovery unit (PACU). Post-operative pain increases the incidence of nausea/vomiting, oxygen requirements and thus, consequently becoming a major barrier to recovery. If found to be effective, post-induction TAP blocks could become the standard of care for regional anesthesia following laparoscopic bariatric surgery and could reduce intra-operative anesthetic and opioid use, opioid consumption in (PACU), post-operative nausea and vomiting and overall length of stay in PACU. This in turn will improve patient's recovery, reduce delays in PACU and decrease patient's length of stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary bariatric surgery at St. Joseph's Healthcare Hamilton surgery including Sleeve Gastrectomy (SG) or Roux-en-Y Gastric Bypass Surgery (RYGB)
* Patients >18 Years of Age

Exclusion Criteria:

* Patients undergoing a revisional bariatric surgery
* Patients with a history of chronic pain or opioid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Immediately post-op
  Opioid Consumption in the post- anesthetic recovery unit

SECONDARY OUTCOMES:
Length of Stay | immediately post-operative
  Length of Stay in post- anesthetic recovery unit
Anesthesia requirements | Intra-operatively
  Intraoperative Anesthesia consumption
Sedation requirements | post-operative up to 24 Hours
  Level of Sedation in Post-operative recovery unit
Nausea and vomiting | post-operative up to 24 Hours
  Incidence of post operative nausea and vomiting
Respiratory Status | immediately post-operative
  Respiratory Status in Post-operative Recovery Unit
Opioid consumption | 24 hours post-operative
  Opioid consumption in the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton - Charlton Campus, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No